CLINICAL TRIAL: NCT07061847
Title: Bilateral Middle Meningeal Artery Lidocaine Infusion for Chronic Debilitating Migraines
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Jeffrey Katz, Principal Investigator, Northwell Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB #: 24-0279
Record Dates: First submitted 2025-07-01; First posted 2025-07-11 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Migraine
Keywords: migraine; headache; intervention; lidocaine; endovascular
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — Lidocaine; Pharmaceutical Preparations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lidocaine (Experimental): All patients who meet eligilibity criteria at their baseline visit will be scheduled for the Lidocaine procedure.
  Interventions: Drug: Lidocaine (drug); Procedure: Lidocaine Procedure

INTERVENTIONS:
Drug: Lidocaine (drug) — The study intervention involves the use of 1% cardiac preservative-free lidocaine. Lidocaine is a local anesthetic commonly used in medical procedures to numb a specific area of the body. In this case, the lidocaine is formulated at a concentration of 1% and will be diluted to 50 mL with normal saline.
  This treatment is an intra-arterial bilateral lidocaine infusion into the middle meningeal artery (i.e. this is a lidocaine infusion into the brain blood vessels to turn off the pain receptors responsible for causing chronic headaches). Lidocaine is an FDA approved anesthetic (i.e. pain killer) used in common medical practice. Lidocaine, however, has not yet been approved by the FDA for this particular use. For this reason, the use of lidocaine in this study is considered investigational.
Procedure: Lidocaine Procedure — All patient who meet eligibility criteria at their baseline visit will be scheduled for the Liocaine procedure.

SUMMARY:
The main purpose of this study is to evaluate the effectiveness of a new treatment in improving chronic migraine symptoms. This treatment involves a targeted lidocaine infusion into blood vessels in the skull to numb pain receptors, potentially leading to improvements in chronic migraine intensity, frequency, and duration.

DETAILED DESCRIPTION:
Given the current literature and using intent-to-treat clinical judgement, the research team believes that the treatment offered in this study may offer a promising benefit to treatment resistant migraine patients. Despite modest advances in drug therapy, some patients still suffer from chronic migraines. Therefore, the headache medicine community continues to search for alternative treatments in the form of research.

The research team is conducting a prospective observational study to gather data before and after this treatment is administered to determine whether there is improvement in migraine duration, intensity, and frequency.

This treatment is an intra-arterial bilateral lidocaine infusion into the middle meningeal artery (i.e. this is a lidocaine infusion into the brain blood vessels to turn off the pain receptors responsible for causing chronic headaches).

Lidocaine is an FDA approved anesthetic (i.e. pain killer) used in common medical practice. Lidocaine, however, has not yet been approved by the FDA for this particular use. For this reason, the use of lidocaine in this study is considered investigational.

This is NOT the first time this procedure has been performed. Intra-arterial lidocaine infusion has been used safely during the treatment of other brain diseases. Infusing brain vessels with lidocaine is not new technique. The treatment offered in this study is new for the treatment of migraines. This particular treatment has been performed successfully in the small group studies that the study investigators are modeling after. The investigative neuro-interventionists have been rigorously trained for this approach and hold a minimum of double board certifications. This team is experienced in using these techniques for other brain diseases and have successfully performed this specific procedure in a select group of early patients. Collectively, the team holds over 45+ years of experience in performing neuro-endovascular procedures.

During the intra-arterial infusion of lidocaine for treatment of a subdural procedure, an incidental finding noted that patients had reduced headache intensity following this treatment.

Therefore, this technique has been re-purposed in this study to treat chronic migraine sufferers. The procedure is considered investigational because lidocaine is not yet FDA-approved for this specific use. Although several studies have demonstrated that this approach is a safe and tolerable treatment for chronic migraine, there is still insufficient evidence to incorporate it into the current day standard of care protocol.

Ultimately, the purpose of this study is to explore this approach to and determine if this treatment can induce a significant improvement in chronic migraine, intensity, duration, and frequency.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 to 75 years with a very severe to extremely severe medically refractory Chronic Daily Headache (CDH).

   1. Chronic: as defined by the International Headache Society Classification ICHD 3 (>15 headache days a month for a period of at least 3 months)
   2. Medically refractory: defined as failure of ≥3 headache preventative treatments.
   3. Severely disabling (Migraine Disability Assessment [MIDAS] Tool score of ≥ 21 [Grade IV])
   4. Score of 6 (very severe) or 7 (extremely severe) on the Global Assessment of Migraine Severity (GAMS) rating scale.
   5. Head pain is at least moderate-to-severe intensity (>5 on a Visual Analog Scale) in ≥50% of headaches.
2. Diagnosis of CDH for ≥ 12 months before screening based on medical records and/or patient self-report.
3. Headache frequency: minimum 15 monthly headache days (MHD) on average across the 3 months prior to screening
4. Patient reports to their provider intolerance or insufficient response with their current preventive treatment (i.e. insufficient reduction in headache frequency, duration, and severity on a standard treatment on a generally accept therapeutic dose for 6 weeks).
5. On a stable concomitant medication and headache preventive for the 3 months prior to screening

During Baseline Period:

1. Must have ≥ 15 MHD based on the patient self-maintained diary data during the baseline period.
2. Must have demonstrated >75% compliance with diary data for the 28 day duration period, or longer if their baseline period carries on past this point.
3. Must continue to meet eligibility criteria when reassessed at baseline completion visit

Exclusion Criteria:

1. Recently started new migraine preventative treatment regimen within the past 3 months.
2. Known allergy or sensitivity to lidocaine.
3. Lidoderm patch (not an exclusion if the Lidoderm patch has been removed for ≥ 3 days before the procedure)
4. Severe allergy/anaphylaxis to iodinated contrast dye.
5. Any intracranial pathology on brain imaging (head CT or MRI within the past 12 months)
6. Chronic subdural hematoma
7. Ischemic stroke or myocardial infarction within 3 months 8. History of renal insufficiency with Cr > 1.5 within 3 months (will be retested during pre-surgical

testing).

9. History of abnormal ECGs within 3 months, specifically:

1. Prolonged QT syndrome
2. Use of medications that may prolong the QT interval such as: anti-nausea, anti-emetics, etc.

   10. Taking any antiarrhythmic medication (other than a beta blocker)

   11. Symptomatic peripheral arterial disease

   12. Known inherited or acquired bleeding diathesis (not including antiplatelet or anticoagulation medication)

   13. Evidence of active substance-related disorders, addictive disorders, or "recreational use" of illicit drugs.

a. If any of these disorders have occurred within 12 months prior to screening, based on medical records, patient self-report, or positive urine drug test (except for prescribed medications that may result in a positive urine drug test).

14. Active chronic pain syndromes (e.g., fibromyalgia and chronic pelvic pain).

15. History of major psychiatric disorder or current evidence of moderately severe or severe depression based on a Patient Health Questionnaire-9 (PHQ-9) total score ≥ 15 at screening.

a. Subjects with history of anxiety disorder and/or major depressive disorder with PHQ-9 < 15) and are taking no more than 1 medication, for each disorder, for at least 2 months prior to screening may be considered.

16. If the subject is pregnant, planning on pregnancy during the duration of the study, or planning on making their partner pregnant will be excluded from the study unless proper contraception is in place.

17. Any diagnosis at the discretion of the investigator that would make the patient unfit.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2027-03-10 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Reduction in Monthly Migraine Headache Days | From enrollment to post-treatment at 3 months
  To observe a ≥50% reduction in monthly migraine headache days in one month post intra-arterial lidocaine infusion into the bilateral middle meningeal artery.

SECONDARY OUTCOMES:
≥50% reduction in migraine headache intensity at 15 minutes, 2 hours, and 24 hours post procedure. | 15 minutes, 2 hours, and 24 hours post-procedure.
Sustained freedom from headache pain >48hrs. | >48hrs post treatment
Percentage of patients achieving ≥75% and 100% reduction in monthly headache days at 1 month and 3 months | At 1 month and 3 month post procedure
Mean number of monthly migraine headaches days at 1 month and 3 months. | From enrollment to 1 month and 3 months post procedure
Mean change from baseline in the Global Assessment of Migraine Severity (GAMS) at 3 months | From enrollment to 3 months post procedure
Percent with improvement in Migraine Disability Assessment (MIDAS) at 3 months from severe disability (Grade IV, score ≥21) to no moderate disability (Grade I to III, score 0-21) | From enrollment to 3 month post procedure
Percent Headache Impact Test (HIT)-6 score <50 at 3 months. | From enrollment to 3 months post procedure
Percent with reduction in need for analgesic use by ≥50% at 3 months. | From enrollment to 3 months post procedure
Adverse events at 24 hours and 3 months post-procedure. | From enrolllment to 3 months post procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Neuroscience Institute at Great Neck, Great Neck, New York, United States

IPD SHARING:
Plan to Share IPD: No